CLINICAL TRIAL: NCT05735626
Title: Treatment of Acute Post-stroke Oropharyngeal Dysphagia With Paired Stimulation Through Peripheral TRVP1 Agonists and Non-invasive Brain Stimulation
Brief Title: Treatment of Acute Post-stroke Oropharyngeal Dysphagia With Paired Stimulation
Acronym: ICI20/00117
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Collaborators: Consorci Sanitari del Maresme (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Pere Clave, Director of Research and Academic Development at CSdM, Hospital de Mataró
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STROD_ICI_A
Record Dates: First submitted 2023-01-17; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Stroke, Acute; Oropharyngeal Dysphagia; Swallowing Disorder
Keywords: TRPV1 agonists; TRPV1/A1 agonists; Transcranial Direct Current Stimulation; Non-invasive Brain Stimulation; Sensory Stimulation; Capsaicin
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — piperine; Capsaicin

STUDY DESIGN:
Intervention Model Description: 2 days randomized crossover study with 60 patients in 3 treatment groups:
  * Piperine 150μM + tDCS 2mA 20'
  * Piperine 1mM+ tDCS 2mA 20'
  * Capsaicin 10μM + tDCS 2mA 20
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding will be applicable for clinical and instrumental assessments for investigators, and for intervention condition for patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piperine 150μM + tDCS 2mA (Experimental): tDCS will be applied for 20 minutes at 2.0 mA (NeuroConn, Germany) with the anode electrode positioned over the pharyngeal primary motor cortex (M1) of the unaffected hemisphere (3.5 cm lateral / 1 cm anterior to the vertex) and the cathode over the opposite supraorbital region. During central stimulation, 5 ml of piperine (150μM) will be administered orally every 5 min. After each administration, the patient will be asked to perform dry swallows every minute. In order to avoid alterations in the safety and efficacy of swallowing during the procedure, the bolus will be rheologically adapted according to the patient's requirements.
  Crossover study, each arm includes a placebo + sham stimulation in one of the two days of treatment. Patients will initiate either placebo + sham stimulation or piperine + tDCS randomly in the first or second day depending on the randomization.
  Interventions: Combination Product: Piperine 150μM + tDCS 2mA
- Piperine 1mM+ tDCS 2mA (Experimental): tDCS will be applied for 20 minutes at 2.0 mA with the anode electrode positioned over the pharyngeal primary motor cortex (M1) of the unaffected hemisphere (3.5 cm lateral / 1 cm anterior to the vertex) and the cathode over the opposite supraorbital region. During central stimulation, 5 ml of piperine (1 mM) will be administered orally every 5 min. After each administration, the patient will be asked to perform dry swallows every minute. In order to avoid alterations in the safety and efficacy of swallowing during the procedure, the bolus will be rheologically adapted according to the patient's requirements.
  Crossover study, each arm includes a placebo + sham stimulation in one of the two days of treatment. Patients will initiate either placebo + sham stimulation or piperine + tDCS randomly in the first or second day depending on the randomization.
  Interventions: Combination Product: Piperine 1mM + tDCS 2mA
- Capsaicin 10μM + tDCS 2mA (Experimental): tDCS will be applied for 20 minutes at 2.0 mA with the anode electrode positioned over the pharyngeal primary motor cortex (M1) of the unaffected hemisphere (3.5 cm lateral / 1 cm anterior to the vertex) and the cathode over the opposite supraorbital region. During central stimulation, 5 ml of capsaicin (10 μM) will be administered orally every 5 min. After each administration, the patient will be asked to perform dry swallows every minute. In order to avoid alterations in the safety and efficacy of swallowing during the procedure, the bolus will be rheologically adapted according to the patient's requirements.
  Crossover study, each arm includes a placebo + sham stimulation in one of the two days of treatment. Patients will initiate either placebo + sham stimulation or capsaicin + tDCS randomly in the first or second day depending on the randomization.
  Interventions: Combination Product: Capsaicin 10μM + tDCS 2mA

INTERVENTIONS:
Combination Product: Piperine 150μM + tDCS 2mA — 2 days treatment with either sham + placebo or piperine 150μM + tDCS 2mA (cross-over randomized study).
  Arms: Piperine 150μM + tDCS 2mA
Combination Product: Piperine 1mM + tDCS 2mA — 2 days treatment with either sham + placebo or piperine 1mM + tDCS 2mA (cross-over randomized study).
  Arms: Piperine 1mM+ tDCS 2mA
Combination Product: Capsaicin 10μM + tDCS 2mA — 2 days treatment with either sham + placebo or capsaicin 10μM + tDCS 2mA (cross-over randomized study).
  Arms: Capsaicin 10μM + tDCS 2mA

SUMMARY:
According WHO, oropharyngeal dysphagia (OD) is a prevalent post-stroke (PS) condition involving the digestive system (ICD-10: I69.391) and an independent risk factor for malnutrition and pulmonary infection; and leads to greater morbimortality and healthcare costs and poorer quality of life (QoL). Currently, OD therapy is mainly compensatory, with low rates of compliance and small benefit, and there is no pharmacological treatment, so new treatments that improve patients' condition are crucial. PS-OD patients present both oropharyngeal sensory and motor deficits, so neurorehabilitation treatments which target both could be optimum. Benefits of paired peripheral sensory stimulation with oral capsaicin or piperine and of central motor noninvasive brain stimulation techniques such as transcranial direct current stimulation (tDCS) will be studied. Pairing sensory peripheral and central stimulation may produce greater benefits. The main aim of the project is to study the efficacy of a novel protocol of paired stimulation on acute PS-OD patients. The investigators will assess the acute application of tDCS/piperine or tDCS/capsaicin in the acute phase of stroke, will improve PS-OD. 2 days randomized crossover study with 60 patients in 3 treatment groups (60 patients in the acute stroke phase divided in 3 study arms). We will assess changes in swallow safety, and neurophysiology of the swallow, hospital stay, respiratory and nutritional complications, mortality and QoL.

DETAILED DESCRIPTION:
* Main hypothesis: Paired neurorehabilitation treatment targeting both pharyngeal sensory and motor components simultaneously through a peripheral pharmacological stimulant (transient receptor potential cation channel [TRPV1] agonist, capsaicin) and central stimulation (NIBS) (tDCS) can improve swallowing function in acute PS-OD patients by promoting cortical plasticity, their QoL and reduce OD associated complications.
* Main objectives: to study the efficacy of a novel protocol of paired stimulation on acute PS-OD patients. The investigators will assess the acute application of tDCS/piperine or tDCS/capsaicin in the acute phase of stroke.
* Secondary aims: to assess 1) safety and adverse events; 2) the effects on safety of swallow with a standardized protocol of swallowing evaluation; 3) clinical outcomes at 3 months follow up; 4) the effect of the treatments on spontaneous swallowing frequency and responsiveness to treatment according to stroke characteristics; 5) the effect in the acute phase on functional severity of OD and specific clinical outcomes.
* Design: 2 days randomized crossover study with 60 patients in 3 treatment groups (60 patients in the acute stroke phase divided in 3 study arms). We will assess changes in swallow safety, and neurophysiology of the swallow, hospital stay, respiratory and nutritional complications, mortality and QoL.
* Study population: 60 Acute PS-OD hospitalized patients.
* Inclusion criteria: Adult patients consecutively admitted with recent (<1month) unilateral hemispheric stroke; impaired safety of swallow (ISS) (V-VST); conscious (NIHSS quest. 1a=0); able to follow the protocol and to give written informed consent (WIC).
* Exclusion criteria: Pregnancy; life expectancy <3m or palliative care; neurodegenerative disorder or previous OD; implanted electronic device; epilepsy; metal in the head; participation in another clinical trial in the previous month.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral acute stroke (up to 15 days of evolution).
* Impaired safety or efficacy of swallow according the volume-viscosity swallowing test (V-VST).
* Conscious patient (NIHSS 1a = 0).
* Patient able to follow the protocol and give written informed consent or, failing that, by a family member or legal representative.

Exclusion Criteria:

* Pregnancy.
* Life expectancy less than 3m or palliative care.
* Neurodegenerative disorder.
* Comprehension aphasia.
* Dementia (GDS 4 or higher).
* Previously diagnosed oropharyngeal dysphagia (dysphagia not related to stroke).
* Implanted electronic device.
* Epilepsy.
* Metal in the head.
* Patients with suspected or PCR-confirmed SARS-CoV-2 infection
* Participation in another clinical trial in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Changes in swallowing function | Day 1, +24 hours, and at 3 months follow-up.
  Changes in the volume-viscosity swallowing test to assess prevalence of signs of impaired efficacy and safety of swallow. Evaluated at visit baseline, post-treatment and at 3 months follow-up).
Changes in spontaneous swallowing frequency | Day 1, +24 hours, and at 3 months follow-up.
  Changes in the electromyographical evaluation of spontaneous swallowing frequency obtaining the number of swallows/min, the amplitude and the latency of swallows. 5 times pre-post treatment visits 1 and pre-post treatment visit 2 and 1 time at 3 months follow-up.

SECONDARY OUTCOMES:
Nutritional status (MNA-sf) | Baseline and 3 months follow-up visits.
  Mini nutritional assessment short form score (nutritional status questionnaire).
Anthropometrics | Baseline and 3 months follow-up visits.
  Weight, height and body mass index.
Bioimpedance | Day 1, +24 hours, and at 3 months follow-up.
  Bioimpedance parameters (total body water, extracellular water, intracellular water, phase angle, muscle mass and cell mass)
Blood analysis | Baseline and 3 months follow-up visits.
  Analytical parameters (albumin, pre-albumin, total protein, total lymphocytes and total cholesterol).
Neuropeptides in saliva determination | Day 1, +24 hours, and at 3 months follow-up.
  Determination by ELISA of concentration of the neuropeptides substance P and CGRP (Calcitonin gene-related peptide) in saliva sample.
Length of hospital stay | From baseline to the end of the study (3-months follow-up visit).
  length of stay during the study.
Aspiration pneumonia admissions | From baseline to the end of the study (3-months follow-up visit).
  Aspiration pneumonia admissions during the study period.
General hospital readmissions | From baseline to the end of the study (3-months follow-up visit).
  General hospital readmissions by any cause during the study period.
Mortality over the study period | From baseline to the end of the study (3-months follow-up visit).
  Mortality over the study period.
Safety of the treatment | From baseline to the end of the study (3-months follow-up visit).
  Safety of the treatment applied (adverse events rate) during all the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, PhD, Principal Investigator — Consorci Sanitari del Maresme
Locations (1):
- Hospital de Mataró. Consorci Sanitari del Mareme., Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Result] Hamdy S, Aziz Q, Rothwell JC, Crone R, Hughes D, Tallis RC, Thompson DG. Explaining oropharyngeal dysphagia after unilateral hemispheric stroke. Lancet. 1997 Sep 6;350(9079):686-92. doi: 10.1016/S0140-6736(97)02068-0. PMID 9291902
- [Result] Cabib C, Ortega O, Kumru H, Palomeras E, Vilardell N, Alvarez-Berdugo D, Muriana D, Rofes L, Terre R, Mearin F, Clave P. Neurorehabilitation strategies for poststroke oropharyngeal dysphagia: from compensation to the recovery of swallowing function. Ann N Y Acad Sci. 2016 Sep;1380(1):121-138. doi: 10.1111/nyas.13135. Epub 2016 Jul 11. PMID 27398981
- [Result] Kumar S, Wagner CW, Frayne C, Zhu L, Selim M, Feng W, Schlaug G. Noninvasive brain stimulation may improve stroke-related dysphagia: a pilot study. Stroke. 2011 Apr;42(4):1035-40. doi: 10.1161/STROKEAHA.110.602128. Epub 2011 Mar 24. PMID 21441148
- [Result] Tomsen N, Ortega O, Alvarez-Berdugo D, Rofes L, Clave P. A Comparative Study on the Effect of Acute Pharyngeal Stimulation with TRP Agonists on the Biomechanics and Neurophysiology of Swallow Response in Patients with Oropharyngeal Dysphagia. Int J Mol Sci. 2022 Sep 15;23(18):10773. doi: 10.3390/ijms231810773. PMID 36142680
- [Result] Wang Z, Wu L, Fang Q, Shen M, Zhang L, Liu X. Effects of capsaicin on swallowing function in stroke patients with dysphagia: A randomized controlled trial. J Stroke Cerebrovasc Dis. 2019 Jun;28(6):1744-1751. doi: 10.1016/j.jstrokecerebrovasdis.2019.02.008. Epub 2019 Apr 5. PMID 30956054
- [Result] Rofes L, Arreola V, Martin A, Clave P. Effect of oral piperine on the swallow response of patients with oropharyngeal dysphagia. J Gastroenterol. 2014 Dec;49(12):1517-23. doi: 10.1007/s00535-013-0920-0. Epub 2013 Dec 11. PMID 24326980
- [Result] Nascimento W, Tomsen N, Acedo S, Campos-Alcantara C, Cabib C, Alvarez-Larruy M, Clave P. Effect of Aging, Gender and Sensory Stimulation of TRPV1 Receptors with Capsaicin on Spontaneous Swallowing Frequency in Patients with Oropharyngeal Dysphagia: A Proof-of-Concept Study. Diagnostics (Basel). 2021 Mar 7;11(3):461. doi: 10.3390/diagnostics11030461. PMID 33799960
- [Result] Alvarez-Larruy M, Tomsen N, Guanyabens N, Palomeras E, Clave P, Nascimento W. Spontaneous Swallowing Frequency in Post-Stroke Patients with and Without Oropharyngeal Dysphagia: An Observational Study. Dysphagia. 2023 Feb;38(1):200-210. doi: 10.1007/s00455-022-10451-3. Epub 2022 Apr 23. PMID 35460440